CLINICAL TRIAL: NCT06055114
Title: Study on Vaginal Microecology and Cervical Local Immune Function in Patients With Uterine Fibroids of Childbearing Age
Status: Not yet recruiting | Type: Observational
Sponsor: Lin Yuan (Other)
Responsible Party: Sponsor-Investigator, Lin Yuan, technologist in charge, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: qfsjyk15853128210
Record Dates: First submitted 2023-09-10; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Uterine Fibroids
Keywords: uterine fibroids; vaginal microecology; cervical local immune function; childbearing age
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Age 20-49 years old; Premenopausal; Clinical diagnosis of uterine myoma; Cervical liquid-based cytology and human papillomavirus typing test are negative.
  Interventions: Diagnostic Test: Microscopic examination of vaginal discharge
- Healthy control group: Age 20-49 years old; Premenopausal; Uterine B-ultrasonography is normal; Cervical liquid-based cytology and human papillomavirus typing test are negative; No vaginal infection.
  Interventions: Diagnostic Test: Microscopic examination of vaginal discharge

INTERVENTIONS:
Diagnostic Test: Microscopic examination of vaginal discharge — Using gram-stained smears to detect vaginal secretions, and then the concentration and diversity of bacterial flora are observed using a microscope.

SUMMARY:
The study participants are patients with uterine fibroids and healthy physical examination subjects from the First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital). The main purpose of this study is to analyze the correlation between uterine fibroids and vaginal microecology and cervical local immune function in patients of childbearing age.

DETAILED DESCRIPTION:
(1) In this study, 150 women of childbearing age who are diagnosed with uterine fibroids in the First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital) are selected as the study group; The differences of vaginal microenvironment and cervical local immune function are compared between 150 healthy women of childbearing age in the same period. (2) After the patients are enrolled, the general information (age, height, weight), menstrual status (age of menarche, menstrual period, cycle, bleeding pattern), clinical manifestations (abnormal uterine bleeding, infertility, abdominal pain), and previous medical history (hypertension, thyroid disease, etc.) of 150 patients with uterine fibroids will be collected. After the end of the first part of the experiment, 150 patients with uterine fibroids will be grouped according to vaginal microecological diagnosis, and the clinical characteristics of patients with uterine fibroids will be analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

Study group inclusion criteria:

* Age 20-49 years old
* Premenopausal
* Clinical diagnosis of uterine myoma
* Cervical liquid-based cytology and human papillomavirus typing test are negative

Healthy control group:

* Age 20-49 years old
* Premenopausal
* Uterine B-ultrasonography is normal
* Cervical liquid-based cytology and human papillomavirus typing test are negative
* No vaginal infection

Exclusion Criteria:

Exclusion criteria of the study group:

* Used antibiotics, hormones, immunosuppressants and regulators within 1 month
* Sex, vaginal irrigation or applied medicine 3 days before the vaginal discharge sampling
* Pregnant, lactating or menstruating women
* Uterus and uterine adnexa have other lesions

Exclusion criteria of healthy control group:

* Used antibiotics, hormones, immunosuppressants and regulators within 1 month
* Sex, vaginal irrigation or applied medicine 3 days before the vaginal discharge sampling
* Pregnant, lactating or menstruating women

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital) examined the uterine fibroid patients and healthy physical examination subjects.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-09 (Estimated)

PRIMARY OUTCOMES:
Bacterial vaginitis (BV) of vaginal microecosystem-150 people in each group | through study completion, an average of 2.5 year
  Nugent score is currently an internationally accepted diagnostic method for BV. Lactobacillus, Gardnerella vaginalis, bacterioid bacteria and campylobacter with variable staining are evaluated by Gram staining and semi-quantitative evaluation method. The total score is the sum of the scores of the above 4 bacteria. 0 to 3 points: normal; 4 ~ 6 points: intermediate BV; ≥7 points: BV

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yuan, Ph.D., Principal Investigator — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The plan will be shared after the clinical trial is completed and the patent protection is obtained

REFERENCES:
- [Result] Yang Q, Ciebiera M, Bariani MV, Ali M, Elkafas H, Boyer TG, Al-Hendy A. Comprehensive Review of Uterine Fibroids: Developmental Origin, Pathogenesis, and Treatment. Endocr Rev. 2022 Jul 13;43(4):678-719. doi: 10.1210/endrev/bnab039. PMID 34741454
- [Result] El Andaloussi A, Chaudhry Z, Al-Hendy A, Ismail N. Uterine Fibroids: Bridging Genomic Defects and Chronic Inflammation. Semin Reprod Med. 2017 Nov;35(6):494-498. doi: 10.1055/s-0037-1607240. Epub 2017 Nov 3. No abstract available. PMID 29100237
- [Result] Zannotti A, Greco S, Pellegrino P, Giantomassi F, Delli Carpini G, Goteri G, Ciavattini A, Ciarmela P. Macrophages and Immune Responses in Uterine Fibroids. Cells. 2021 Apr 22;10(5):982. doi: 10.3390/cells10050982. PMID 33922329